CLINICAL TRIAL: NCT02970409
Title: A Randomized Study to Test Peripheral Venous Catheter Lock Therapy With Either Heparin or Saline in Patients Admitted to the Internal Medicine Department
Brief Title: Heparin Versus Saline in Peripheral Venous Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundación para la Investigación Biomédica del Hospital Gregorio Maranon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIBHGM-ECNC002-2014
Record Dates: First submitted 2015-10-15; First posted 2016-11-22 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- heparin (Active Comparator): Catheter Lock Therapy with Heparin
  Interventions: Device: Heparin
- saline (Experimental): Catheter Lock Therapy with saline
  Interventions: Device: saline

INTERVENTIONS:
Device: saline — catheter lock using saline
  Arms: saline
Device: Heparin — catheter lock using Heparin
  Arms: heparin

SUMMARY:
A clinical, prospective. controlled and randomized study with patients with a peripheral venous catheter. Patients will be randomized to either receive heparin or saline. The investigators will monitored the clinical out come to further evaluate catheter colonization rate, phlebitis rate, days of hospital stay, antimicrobial costs, and adverse effects.

DETAILED DESCRIPTION:
The need of use of peripheral venous catheters and the importance of a proper management to avoid catheter colonization or phlebitis requires two possible preventive approaches: lock therapy with heparin or saline.

Heparin demonstrated its efficacy in central venous catheters, but there are still controversies of whether it is useful in peripheral venous catheters.

Objectives To compare the efficacy of heparin in peripheral venous catheters lock versus saline for the prevention of colonization and phlebitis in patients admitted to an Internal Medicine Department.

Methods: A clinical, prospective. controlled and randomized study with patients with a peripheral venous catheter.

Patients will be randomized to either receive heparin or saline. The investigators will monitored the clinical out come to further evaluate catheter colonization rate, phlebitis rate, days of hospital stay, antimicrobial costs, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* patients with inserted PV Catheter within 24h from admission in internal medicine

Exclusion Criteria:

* hypersensibility to heparin
* active hemorrhage
* coagulation alterations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2015-10-17 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
complications | Daily from catheter insertion until catheter withdraw(estimated 10 days)
  prevention of colonization(superficial and tip culture) and phlebitis(visual inflammation of entrance of catheter insertion) .

SECONDARY OUTCOMES:
catheter related infection rate | Through study completion( estimated 2 year after Last patient in)
  episodes of catheter related infection against number of days of exposure to catheter
adverse events(number of catheter obstructions and coagulation alterations) | Through study completion (2 year afterLast patient in)

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine Department HGU Gregorio Marañón, Madrid, Spain